CLINICAL TRIAL: NCT00566124
Title: No Evidence for Essential Differences Between the Effects of Insulin Glargine, Insulin Detemir and NPH Insulin on Glucose Metabolism After a Single Injection as Assessed by 24-h Euglycemic Clamp Studies in Healthy Humans
Brief Title: Basal Insulins - Pharmacodynamics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Diabetes Association (Other); The Institute of Experimental Clinical Research, University of Aarhus (Unknown); Novo Nordisk A/S (Industry)
Responsible Party: Ole E. Schmitz, DMSc., University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Opus 1; 2004-41-4474; 20040188; 2612-2731
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes
Keywords: Levemir, Lantus, Insulatard, Pharmacodynamics, Healthy humans
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir; Insulin Glargine; Isophane Insulin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Insulin detemir
  Interventions: Drug: Insulin detemir
- 2 (Active Comparator): Insulin glargine
  Interventions: Drug: Insulin glargine
- 3 (Active Comparator): NPH insulin
  Interventions: Drug: Insulatard

INTERVENTIONS:
Drug: Insulin detemir — 0.4 U/kg bw insulin detemir injected s.c. in the thigh.
  Other Names: Levemir
  Arms: 1
Drug: Insulin glargine — 0.4 U/kg bw insulin glargine injected s.c. in the thigh
  Other Names: Lantus
  Arms: 2
Drug: Insulatard — 0.4 U/kg bw NPH insulin injected s.c. in the thigh
  Arms: 3

SUMMARY:
To purpose of this study is to compare the pharmacodynamic properties of insulin detemir, insulin glargine and NPH insulin after a single subcutaneous injection.

DETAILED DESCRIPTION:
In this randomized, double-blind, euglycemic glucose clamp study, 10 healthy male volunteers received a subcutaneous injection of 0.4 U/kg insulin detemir, insulin glargine or NPH insulin on three separate study days in a cross-over design. After insulin administration, plasma glucose was maintained at 0.3 mmol/l below fasting level for 24 hours by manually adjusted glucose infusion. C-peptide, insulin, NEFA and counter regulatory hormones were measured throughout the clamp period. Endogenous glucose release (EGR) was assessed by the isotope dilution technique (3-3H-glucose).

ELIGIBILITY:
Inclusion Criteria:

* Male
* BMI 20 - 50 kg/m2
* Blood pressure < 140/90 mmHg
* signed informed consent
* Caucasien

Exclusion Criteria:

* Diabetes or other disease
* Alcohol or drug abuse
* Smoking
* Use of prescription drugs

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Area under GIR-curve, maximal glucose infusion rate, time to maximal glucose infusion rate. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ole E. Schmitz, DMSc, Principal Investigator — University of Aarhus
Locations (1):
- Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus, DK, Denmark